CLINICAL TRIAL: NCT04921618
Title: Towards Improving Information, Testing and Treatment for Partners of People Diagnosed With STIs in Testing Centres and Sexual Health Clinics, the Not'IST Study
Brief Title: Partner Notification of Sexually Transmitted Infections (STIs) in Testing Centers
Acronym: Not'IST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS MIE Not'IST
Record Dates: First submitted 2021-04-27; First posted 2021-06-10 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: STI; Hiv
Keywords: partner notification; STI; HIV; testing center; intervention design
MeSH Terms: conditions — Sexually Transmitted Diseases; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Index patients: People aged 18 or more diagnosed with >= 1 STI in testing centers.
  [STI = bacterial STIs and/or HIV and/or acute hepatitis C virus (HCV)]
  Interventions: Other: 2 online self-administered questionnaires on
- Notified partners: People aged 18 or more getting STI testing in testing centers after being notified by a sexual partner.
  [STI = bacterial STIs and/or HIV and/or acute HCV]
  Interventions: Other: 2 online self-administered questionnaires on

INTERVENTIONS:
Other: 2 online self-administered questionnaires on — 1. Participant profile
  2. Spontaneous partner notification practices collected one month after STIs diagnosis
  Groups: Index patients
Other: 2 online self-administered questionnaires on — 1. Participant profile
  2. Experiences with partner notification and use of STI testing following notification
  Groups: Notified partners

SUMMARY:
Since the 2000s, the incidence of bacterial STIs increases, mainly among men who have sex with men but also among heterosexual men and women with multiple sexual partners. A partner notification (PN) approach could break transmission chains and curb STI epidemics. PN brings together a set of interventions to help people diagnosed with STIs to inform their partners, encourage them to get tested, so that they can access treatment or prevention. A PN approach, systematically offered at STI diagnosis, has not yet been implemented in France and needs to be evaluated. In 2018, the Conseil National du Sida (French National AIDS Council) stated in favor of a formalized PN approach, particularly in testing centers, which carry out a large part of STI diagnoses.

The aim of our research project is to build interventions facilitating information, testing and treatment of partners of people diagnosed with STIs in testing centers and sexual health clinics.

Step 1: A cross-sectional study

Primary objective

To describe the PN practices of people diagnosed with an STI in testing centers and sexual health clinics without any intervention

Secondary objectives

* To describe the profiles of people diagnosed with an STI in testing centers or sexual health clinics and therefore likely to receive an intervention to help them notify their partners;
* To describe the profiles of people notified by their partners and who attend testing centers or sexual health clinics for STI testing;
* To describe the notification received by these notified partners and identify the facilitators of testing use following notification.

Step 2: A qualitative study

Objectives

* To evaluate the acceptability of testing center staff for an STI notification program in general and discuss the feasibility of interventions pre-identified by a literature review;
* In a collaborative (researchers and staffs) approach, to adapt these interventions to (1) the testing centers working and (2) the needs of their users identified in the cross-sectional study.

Expected results

This study is the first step in implementation of a PN program as part of a comprehensive management of STI diagnoses in France.

DETAILED DESCRIPTION:
Methods

Step 1: A cross-sectional study

Cross-sectional study conducted in testing centers and sexual health clinics (6 centers, 6 months of enrollment), targeting two populations:

* People aged 18 years or more diagnosed for at least one STI: the index patients;
* People aged 18 years or more attending the same centers for STI testing after being notified by a sexual partner: the notified partners.

This study is based on 3 online self-administered questionnaires:

* A questionnaire, the same for index patients and notified partners, collecting socio-demographic profile, health care and testing use, STI history and sexual behavior;
* A questionnaire for index patient on spontaneous PN practices of index patients one month after STI diagnosis, including types of partners notified, methods used to notify, and reasons for not notifying partners (this questionnaire will be sent one month after STI diagnosis to give participants the time to inform their partners);
* A questionnaire for notified partner on their experience of PN, such as the type of notifying partner, the methods and information transmitted during notification, their feelings and what led them to get testing after being notified.

A notified partner diagnosed with an STI will receive also the questionnaire on spontaneous practices of index patients at M1. This will allow us to observe whether people who had already been notified for an STI are more likely to notify their partners.

Step 2: A qualitative study

Focus-groups of 6-8 volunteers involved in STI testing in testing centers and sexual health clinics will be conducted based on an interview guide. Doctors and other staffs will be interviewed separately.

Thematic analysis

ELIGIBILITY:
Inclusion Criteria:

For index patients

* Diagnosed with at least one bacterial STI, and/or HIV and/or acute HCV at one of the participating centers during the study period,
* Aged >= 18,
* Agree to participate in the study after oral and written information.

For notified partners

* Attend one of the participating centers during the study period, within 6 months of being notified of their exposure to an STI (bacterial STI, and/or HIV and/or acute HCV) by one of their partners, who is infected with one or more of these STIs,
* Aged >= 18,
* Agree to participate in the study after oral and written information.

Non-Inclusion Criteria:

For index patients and notified partners

* People who do not read or speak French,
* Wardship or curatorship adults.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Two distinct populations will be studied
  * People diagnosed with >= 1 STI in testing centers or sexual health clinics: index patients,
  * People attenting testing centers or sexual health clinics for STI testing and/or access to treatment following notification of possible exposure to an STI by one of their partners: notified partners.
  Index patients and notified partners will be included on a voluntary basis. The study will be offered to all eligible individuals during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Partner notification by index patients | One month after STI diagnosis
  Proportion of index patients who notified at least one sexual partner one month after their STI diagnosis

SECONDARY OUTCOMES:
Partners notified by index patients | One month after STI diagnosis
  Mean proportion of notified partners among partners reported by index patients
Notified partners tested positive | At notified partners inclusion
  Proportion of notified partners tested positive among notified partners attending STI testing

CONTACTS AND LOCATIONS:
Overall Officials: Jade Ghosn, Pr, Principal Investigator — IAME, Inserm UMR1137, Paris and Infectious diseases department, Bichat Hospital, Paris; Karen Champenois, Principal Investigator — IAME, Inserm UMR1137, Paris
Locations (9):
- France (9):
  - CeGIDD d'Aix-en-Provence, Aix-en-Provence
  - CeGIDD de Caen, Caen
  - CeGIDD de Lille, Lille
  - CeGIDD - La Joliette, Marseille
  - CeGIDD - Saint Adrien, Marseille
  - CeGIDD de Bichât, Paris
  - CeGIDD de La Pitié Salpêtrière, Paris
  - Centre de santé sexuelle - LE 190, Paris
  - Institut Alfred Fournier, Paris